CLINICAL TRIAL: NCT01636570
Title: Double-Blind, Placebo-Controlled Trial of Vitamin D3 (Cholecalciferol) Supplementation for Heart Failure Patients
Brief Title: Vitamin D3 Supplementation for Heart Failure Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidi Moretti, MS, RD (Other)
Collaborators: Saint Patrick Hospital (Other)
Responsible Party: Sponsor-Investigator, Heidi Moretti, MS, RD, Co-Investigator, Saint Patrick Hospital
Organization: Saint Patrick Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VitD3HF
Record Dates: First submitted 2012-07-03; First posted 2012-07-10 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Heart Failure; Vitamin D Deficiency; Cardiomyopathy; Congestive Heart Failure
Keywords: Vitamin D; Cholecalciferol; Heart Failure; Congestive heart failure; Cardiomyopathy; Strength; Parathyroid Hormone; Calcium; Quality of Life; C reactive protein; Cardiopulmonary exercise testing; Prognosis
MeSH Terms: conditions — Heart Failure; Vitamin D Deficiency; Cardiomyopathies | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (cholecalciferol) (Active Comparator): 10,000 International Units of vitamin D3 will be given daily for 6 months in vitamin D deficient heart failure patients.
  Interventions: Drug: Vitamin D3 (cholecalciferol)
- Sugar Pill (Placebo Comparator): Patients will be given an placebo that is identical in appearance to the active comparator. It will be given as 2 gelcaps per day.
  Interventions: Drug: Placebo Comparator: Sugar Pill

INTERVENTIONS:
Drug: Placebo Comparator: Sugar Pill — Placebo will be given in identical gelcaps (as microcrystalline cellulose) as 2 per day for a period of 6 months.
  Other Names: Bio-tech Pharmacal
  Arms: Sugar Pill
Drug: Vitamin D3 (cholecalciferol) — 10,000 IU vitamin D3 will be given as 5000 IU gelcaps two per day for a period of 6 months.
  Other Names: Bio-tech Pharmacal
  Arms: Vitamin D3 (cholecalciferol)

SUMMARY:
The purpose of this study is to determine if treatment with vitamin D3 of 10,000 International Units (IU) daily in vitamin D deficient patients for 6 months will improve B type natriuretic peptide (BNP), a marker of heart function, compared to placebo. The investigators also aim to determine if vitamin D helps cardiopulmonary function as evaluated by cardiopulmonary exercise test (CPX), laboratory values, strength, and quality of life in patients with stable congestive heart failure (Class II or III).

ELIGIBILITY:
Inclusion Criteria:

* NYHA Heart Failure Class II or II, stable
* Vitamin D deficiency (32 ng/ml or less)
* No recent medication changes for 3 months
* Females of childbearing age must use effective contraceptive if they are sexually active

Exclusion Criteria:

* Hypercalcemia
* Nephrolithiases
* Sarcoidosis
* Acute cardiac insufficiency
* Pregnancy
* Breastfeeding
* Any clinically unstable medical condition
* Supplements of greater than or equal to 1000 units of vitamin D per day

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
B type Natriuretic Peptide (BNP) | Change in BNP will be measured at baseline and after 6 months of treatment with vitamin D or placebo
  BNP is a hormone secreted by the heart ventricles, and high concentrations of this hormone occur in heart failure. It is a strong prognostic indicator.

SECONDARY OUTCOMES:
Cardiopulmonary exercise test (CPX) | Change in CPX will be measured at baseline and after 6 months of treatment with Vitamin D3 or placebo
  Secondary outcome measure will include improvements from baseline in cardiopulmonary function as evaluated by CPX(includes measurement of the change in ventilator efficiency (VE/VCO2), partial pressure of end-tidal CO2 (PETCO2)
25 hydroxyvitamin D [25 (OH)D] | Change in 25 hydroxyvitamin D will be measured at baseline, at 12 weeks, and after 6 months of treatment with vitamin D or placebo
  Patients with vitamin D deficiency as defined by 25(OH)D of less than 32 ng/ml. 25(OH)D is the most accurate measurement for assessment of vitamin D status. However, ideal ranges for serum 25 (OH)D have not been well established. A recent pharmokinetic study conducted by Hollis, et al, found that 25 OHD levels had to exceed 40 ng/ml and sometimes 50 ng/ml, for the parent substrate (cholecalciferol) to be detectable in the blood (Hollis 2007. IF 25(OH)D levels exceed 150 ng/ml, they will be withdrawn from the study to avoid toxicity.
C reactive protein (CRP) | Change in CRP will be measured at baseline and after 6 months of treatment with vitamin D or placebo
  CRP is related to heart failure incidence, and vitamin D seems to be inversely related to CRP levels.
Serum Calcium | Change in serum calcium levels will be measured at baseline, at 12 weeks, and at 6 months of treatment with vitamin D or placebo
  Measurement of serum calcium levels will help to assess safety of vitamin D treatment. If serum calcium becomes elevated, patients will be withdrawn from the clinical trial.
6 minute walk test | Change in the 6 minute walk test will be measured at baseline and at 6 months of treatment with vitamin D or placebo
  The 6 minute walk test is used to measure aerobic activity at baseline and after completion of supplemental vitamin D or placebo. This test is an objective measurement of exercise capacity, and has been shown to be reproducible and a suitable measure for outcome in patients with heart failure (Guyatt). The 6 minute walk test in heart failure patients is strongly associated with vitamin D serum concentrations (p=0.002) and inversely with high sensitivity C reactive protein (hsCRP), an inflammatory marker (p=0.001)
Kansas City Cardiomyopathy Questionnaire | Chang in the KCCQ will be measured at baseline and after 6 months of treatment with vitamin D or placebo
  Measurements of quality of life provide means of measuring prospective benefits of heart failure interventions. The KCCQ is associated with hospitalization and mortality, and is sensitive to changes in heart function with ARB, beta-blocker and ACE inhibitor treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley D Berry, MD, Principal Investigator — International Heart Institute of Montana; Heidi D Moretti, MS, RD, Study Director — Saint Patrick Hospital
Locations (2):
- United States (2):
  - International Heart Institute of Montana, Missoula, Montana
  - Saint Patrick Hosptial, Missoula, Montana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moretti HD, Colucci VJ, Berry BD. Vitamin D3 repletion versus placebo as adjunctive treatment of heart failure patient quality of life and hormonal indices: a randomized, double-blind, placebo-controlled trial. BMC Cardiovasc Disord. 2017 Oct 30;17(1):274. doi: 10.1186/s12872-017-0707-y. PMID 29084522